CLINICAL TRIAL: NCT02370108
Title: The Study of Rest Tremor Suppression by Using Electrical Muscle Stimulation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 483/57
Record Dates: First submitted 2015-01-23; First posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Rest Tremor; Parkinson's Disease
Keywords: electrical muscle stimulation; parkinson's disease; rest tremor; tremor reduction
MeSH Terms: conditions — Tremor; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PD patient (Experimental): Parkinson's disease patients will get the electrical muscle stimulation at the most tremulous hand at 50 Hz frequency, maximal tolerate pulse amplitude (not over 20 mA), duration of stimulation for 10 second.
  Interventions: Device: electrical muscle stimulation
- OT patients (Experimental): others tremor patients will get the electrical muscle stimulation at the most tremulous hand at 50 Hz frequency, maximal tolerate pulse amplitude (not over 20 mA), duration of stimulation for 10 second.
  Interventions: Device: electrical muscle stimulation

INTERVENTIONS:
Device: electrical muscle stimulation — electrical muscle stimulation at hand muscle for reduction tremor

SUMMARY:
This study is aimed to study the safety and feasibility of electrical muscle stimulation (EMS) in suppression of tremor from various causes especially for rest tremor in Parkinson's disease.

DETAILED DESCRIPTION:
Study method as follows:

* All subjects will be provided the information on this research study and informed consent will be sought for every subjects.
* All subjects (30 PD patients and 30 others tremor patients) will be interviewed by a movement disorders specialist or a trained interviewer for their demographic and clinical data.
* All PD patients will be examined for the severity of Parkinson's disease by a movement disorders specialist according the Unified Parkinson's disease Rating Scale (UPDRS), Hoehn and Yahr score, and tremor rating scale, during the 'on period' in order to determine the additional effect of EMS for suppression of tremor. Physical examinations of each patient will be recorded by the video recording for later reviewed.
* All essential tremor and dystonic tremor patients will be examined by a movement disorders specialist for the tremor severity according to the Fahn, Tolosa, Marin Tremor Rating Scale. Physical examinations of each patient will be recorded by the video recording for later reviewed.

All patient will be determined for feasibility to use EMS and safety of EMS. Pain will determined by visual analog scale.

* All patients will be monitored their hand tremor at resting position and postural position. The tremor analysis with accelerometer and gyroscope system (Parkinson Monitor V0.006 Beta) and the surface EMG (Nicolet EDX Viking) will be conducted. The surface EMG electrode will place over thenar muscle of the hand, which is the most predominant sided of tremor, for quantitative measurement and determination of tremor physiology.
* All participants data from surface EMG will be applied to The Matlab™ program (MathWorks Inc.) in order to modify the qualitative signals into quantitative parameters and performing the high-dimensional feature vectors, and later to determine the different efficacy in pulse amplitude of electrical muscle stimulation on feature vectors.
* The electrical muscle stimulation (Intensity™ Twin Stim® III) will be conducted by placement the 2 self-adhesive electrode (size 1.5 inches * 1.5 inches) over thenar muscle and 1st&2nd interrosseous muscle of the hand, which is the most predominant sided of tremor. The EMS will be stimulated PD patients on the rest position, whereas the other tremors patients in both rest position and postural position. The pulse amplitude will be slowly titration until provided the tetanic muscle contraction (motor threshold) without pain (all applied frequency is 50 Hz).
* All of examination will be taken for 30 minutes for each one subject.

Data Collection

* Demographic and clinical data: age, gender, clinical diagnosis, disease's duration and severity score for each subject according to establishing standard rating scale.
* Tremor parameters form Parkinson Monitor V0.006 Beta will be collected in both before and during EMS as 5 parameters: Peak magnitude, RMS, Angle, Frequency, Q
* The pulse amplitude from EMS will be recorded in every titration in order to determine the efficacy of EMS in difference pulse amplitude.
* The surface EMG and acceleration signal in difference pulse amplitude will be extracted and clustered data in order to analyze by using Matlab™, and performed the high-dimensional feature vectors for quantitative interpretation.

Data Analysis The statistical analysis in this study is based from SPSS program version 17. Categorical data will be analyzed for frequency and percentage. Continuous data will be analyzed by mean and standard deviation (SD). Non-parametric study would be preferred if the small sample size or in case of distribution of data do not present as normal distribution (determined by Kolmogorov-Smirnov test). The repeated ANOVA will be used for determined the efficacy of difference pulse amplitude on tremor suppression and the efficacy of EMS in the difference times in follow up periods.

ELIGIBILITY:
Inclusion Criteria:

* For PD patients

  * Adults ≥ 18 years old.
  * Patients with Parkinson's disease diagnosed according to the UKPDSBB criteria with predominantly feature of rest tremor that intractable to medically treatment.
  * Informed consent For other tremor patients
  * Adults ≥ 18 years old.
  * Patients with essential tremor diagnosed according to the TRIG criteria for essential tremor or patients with dystonic tremor diagnosed according to the proposed definition in which their symptoms shared similar trait of medically intractable tremor.
  * Informed consent

Exclusion Criteria:

* For PD patients

  * Patients with a history of cardiac arrhythmia, renal failure, hepatic failure, and pregnancy as well as those who had history of seizure or had the risk for tended to become seizure such as those who had focal brain lesions, encephalitis, and stroke patients.
  * Patients with a history of hand surgery and implanted screws or wires in hand area that supposed to place a surface EMG or EMS, as well as those patients who were implanted for electrical devices such as cardiac pacemaker, pulse generator of deep brain stimulation,and intrathecal baclofen pump.
  * Patients who cannot avoid the medication that may potentiate or attenuate tremor such as antihistamines, benzodiazepine, illicit drugs, and thyroid hormone supplement.

For other tremor patients

* Patients with a history of cardiac arrhythmia, renal failure, hepatic failure, and pregnancy as well as those who had history of seizure or had the risk for tended to become seizure such as those who had focal brain lesions, encephalitis, and stroke patients.
* Patients with a history of hand surgery and implanted screws or wires in hand area that supposed to place a surface EMG or EMS, as well as those patients who were implanted for electrical devices such as cardiac pacemaker, pulse generator of deep brain stimulation, and intrathecal baclofen pump.
* Patients who cannot avoid the medication that may potentiate or attenuate tremor such as antihistamines, benzodiazepine, illicit drugs, and thyroid hormone supplement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-01 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of participant who had tremor suppression determine by reduction of tremor rating scale during electrical muscle stimulation | up to 1 month follow up
  To determine the number of participant with tremor suppression during electrical muscle stimulation

SECONDARY OUTCOMES:
Number of participant who report pain or any adverse events from electrical muscle stimulation | up to 1 month follow up
  To determine number of participant who report pain or adverse events from electrical muscle stimulation
The severity of pain related from electrical muscle stimulation by visual analog scale | intraoperative
  To determine the severity of pain related from electrical muscle stimulation by visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Roongroj Bhidayasiri, MD, FRCP, Study Director — Chulalongkorn University